CLINICAL TRIAL: NCT05954663
Title: Clinical and Hemodynamic Evaluation After Venous Recanalization of Post-thrombotic Iliofemoral Syndromes
Acronym: CHEVROPIS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_1131
Record Dates: First submitted 2023-07-05; First posted 2023-07-20 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Venous Recanalisation
Keywords: Post-thrombotic syndrome; Deep vein thrombosisA; Endovascular recanalization and stenting; Morphological and hemodynamic echodoppler criteria; Venous stent restenosis
MeSH Terms: conditions — Postthrombotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent venous recanalization by angioplasty-stenting: Patients who underwent venous recanalization by angioplasty-stenting for post-thrombotic iliofemoral syndromes from June 2014 to June 2021.
  Interventions: Other: Basic demographic information

INTERVENTIONS:
Other: Basic demographic information — Basic demographic information: age, sex, weight, height, BMI. Comorbidities: history of major bleeding, cardiovascular comorbidities, diabetes mellitus, renal failure, smoking, hormone therapy Anticoagulant and antiplatelet therapy (molecule, duration and indication, before and after intervention) Procedure data: number and type of stents implanted, diameters and lengths, name of stented venous segments Postoperative complications: bleeding complications, pelvic pain, early thrombosis, early pulmonary embolism
  * Clinical examination carried out 1 month after the operation and more than 6 months after the operation
  * Data from the control ultrasound performed 1 month after the operation and more than 6 months after the operation

SUMMARY:
Post-thrombotic syndrome (PTS) is the most common chronic complication of deep vein thrombosis (DVT). The endovascular recanalization and stenting technique has become the gold standard treatment for medically resistant and disabling PTS.

Stent thrombosis is a significant complication of this procedure; the risk factors for thrombosis are poorly understood.

Monitoring the patency of the stent is a key component in maintaining clinical success.

Doppler ultrasound is the first-line diagnostic tool for monitoring patients with venous stents, and has the potential to allow accurate assessment of venous stent obstruction.

Absence of validated morphological and hemodynamic echodoppler criteria for the follow-up of these stents.

• Main objective: Clinical and hemodynamic results of venous recanalisations by stenting in the chronic phase

• Secondary objective (s):

* External validation of hemodynamic criteria proposed in the literature to detect venous stent obstruction
* Risk factors for venous stent restenosis

ELIGIBILITY:
Inclusion Criteria:

- Disabling post-thrombotic syndrome (venous claudication) after at least 6 months of proximal deep vein thrombosis.

Exclusion Criteria:

* Inability to consent
* Age <18 years old
* Life expectancy <3 months
* Incomplete medical records
* Lost in follow up

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with a disabling post-thrombotic syndrome (venous claudication) after at least 6 months of proximal deep vein thrombosis.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 6 first month post intervention
  Villalta score
  * Score ≤ 4: No TPS.
  * Score between 5 and 14: mild TPS.
  * Score between 10-14: moderate TPS.
  * Score ≥ 15 or ulcer present: severe TPS.
Stent patency | 6 first month post intervention
  Analyze of venous patency of each venous segment Maximum peak flow velocity (in centimetres per second) at each venous segment Location of the implanted stents Cranial and caudal extremity Total length Diameter

CONTACTS AND LOCATIONS:
Locations (1):
- Groupement Hospitalier Edouard Herriot, Lyon, France